CLINICAL TRIAL: NCT02472275
Title: Targeting the Prostatic Tumor Microenvironment With PLX3397, a Tumor-Associated Macrophage Inhibitor in Men With Unfavorable Risk Prostate Cancer Undergoing Radiation Therapy and Androgen Deprivation Therapy
Brief Title: PLX3397, Radiation Therapy, and Antihormone Therapy in Treating Patients With Intermediate- or High-Risk Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elisabeth Heath, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-075; NCI-2015-00742 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1501013723; 2014-075 (Other: Wayne State University/Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Stage I Prostate Adenocarcinoma; Stage II Prostate Adenocarcinoma; Stage III Prostate Adenocarcinoma
MeSH Terms: interventions — Androgen Antagonists; pexidartinib; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (PLX3397, radiation therapy, ADT) (Experimental): Patients receive multitargeted tyrosine kinase inhibitor PLX3397 PO BID for 6 months, undergo radiation therapy for 2 months daily (Monday-Friday) beginning at month 3, and undergo ADT with leuprolide acetate, goserelin acetate, or degarelix injections in any month.
  Interventions: Drug: Antiandrogen Therapy; Other: Laboratory Biomarker Analysis; Drug: Multitargeted Tyrosine Kinase Inhibitor PLX3397; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Antiandrogen Therapy — Undergo ADT with leuprolide acetate, goserelin acetate, or degarelix
  Other Names: ADT; Androgen Deprivation Therapy; Anti-androgen Therapy; Anti-androgen Treatment; Antiandrogen Treatment; Hormone Deprivation Therapy; Hormone-Deprivation Therapy
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Multitargeted Tyrosine Kinase Inhibitor PLX3397 — Given PO
  Other Names: PLX3397
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RADIATION; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase I trial studies the side effects and best dose of multitargeted tyrosine kinase inhibitor PLX3397 (PLX3397) when given together with radiation therapy and antihormone therapy in treating patients with prostate cancer that is at intermediate or high risk of spreading. Multitargeted tyrosine kinase inhibitor PLX3397 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth, and may also help the radiation therapy work better. Radiation therapy uses high-energy x-rays to kill tumor cells. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as leuprolide acetate, goserelin acetate, or degarelix, may lessen the amount of androgens made by the body. Giving multitargeted tyrosine kinase inhibitor PLX3397 with radiation therapy and antihormone therapy may be a better treatment for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To conduct a phase I, dose escalation trial with a primary objective of establishing the maximum tolerated dose (MTD) and the dose limiting toxicity (DLT).

SECONDARY OBJECTIVES:

I. To assess the effects of radiation therapy (RT), androgen deprivation therapy (ADT), and PLX3397 (at its MTD) on tumor-associated macrophages (TAMs) in the prostate biopsy after treatment.

OUTLINE: This is a dose-escalation study of multitargeted tyrosine kinase inhibitor PLX3397.

Patients receive multitargeted tyrosine kinase inhibitor PLX3397 orally (PO) twice daily (BID) for 6 months, undergo radiation therapy for 2 months daily (Monday-Friday) beginning at month 3, and undergo ADT with leuprolide acetate, goserelin acetate, or degarelix injections in any month.

After completion of study treatment, patients are followed up at 20-30 days and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of prostate adenocarcinoma
* Must have confirmed viable archival prostate biopsy tissue available as per Section 8.1 (this will be collected for patients going on study after the MTD has been reached
* Intermediate or high risk prostate cancer patients who are candidates for radiation therapy:
* Gleason >7 or
* Clinical or pathological > T2b disease or
* PSA > 10 ng/mL
* No evidence of metastatic disease by clinical and radiological staging
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1
* No standard contraindications to radiation therapy including prior significant radiation therapy, inflammatory bowel disease, irritable bowel syndrome or collagen vascular disease
* Prior history of up to 8 weeks of androgen deprivation therapy defined as lutenizing-hormone releasing hormone (LHRH) or other medical castration therapy prior to registration is acceptable. This will be in addition to the 6 months of ADT on study.
* Life expectancy of at least 3 months
* Adequate hematologic, hepatic, and renal function as defined by:
* Absolute neutrophil count ≥ 1.5 × 109/L
* Hemoglobin > 10 g/dL
* Platelet count ≥ 100 × 109/L
* AST and ALT ≤ upper limit of normal (ULN)
* TBil and DBil ≤ ULN with an exception of patients with confirmed Gilbert's syndrome. For patients with confirmed Gilbert's syndrome, the TBil should be ≤ 1.5 × ULN
* Serum creatinine ≤ 1.5 × ULN
* Must have ability to take oral medication
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Ability to understand and willingness to sign a written informed consent document
* Willingness to be treated with radiation therapy and androgen deprivation Therapy

Exclusion Criteria:

* Investigational drug use within 28 days of the first dose of PLX3397 or concurrently
* At Screening QTcF ≥450 msec
* Patients with serious illnesses, uncontrolled infection, medical conditions, or other medical history including abnormal laboratory results, which in the investigator's opinion would be likely to interfere with a patient's participation in the study, or with the interpretation of the results
* Refractory nausea and vomiting, malabsorption, biliary shunt, or significant bowel resection that would preclude adequate absorption of study drug
* Known active or chronic human immunodeficiency virus (HIV) or hepatitis C virus (HCV) infection, or positive hepatitis B (Hep B) surface antigen. Prior hepatitis infection that has been treated with highly effective therapy with no evidence of residual infection and with normal liver function (ALT, AST, total and direct bilirubin ≤ ULN) is allowed.
* Hepatobiliary diseases including biliary tract diseases, autoimmune hepatitis, inflammation, fibrosis, cirrhosis of liver caused by viral, alcohol, or genetic reasons. Gilbert's disease is allowed if TBil is ≤ 1.5 × ULN.
* Active cancer (either concurrent or within the last 3 years) that requires nonsurgical therapy (e.g. chemotherapy or radiation therapy), with the exception of surgically treated basal or squamous cell carcinoma of the skin, or melanoma insitu.
* AST/ALT > 2.5X ULN or >5X ULN in the presence of liver metastases.
* Current treatment with anti-androgen is allowed for a maximum of one month to prevent flare response with ADT
* Concomitant use of acid reducing agents (e.g., proton pump inhibitors, H2 receptor antagonists, antacids)
* Concomitant use of strong and moderate CYP3A4 inhibitors and inducers
* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of the study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-06; Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Grade of specific types of toxicity | Up to 30 days after end of study treatment
  Frequency distributions will be generated by dose level, and overall.
MTD of multitargeted tyrosine kinase inhibitor PLX3397, determined according to incidence of DLT | 4 months

SECONDARY OUTCOMES:
Change in metabolic syndrome parameters | Baseline to month 7
  Descriptive statistics will be used to summarize the 7 metabolic syndrome parameters), and changes in them. These statistics will be calculated only for patients treated at the MTD, where the correlatives are measured, and will be generated for all 12 MTD patients combined, and separately by MTD randomization arm.
Change in PSA levels | Baseline to up to month 7
  PSA levels (and their change) will be tabulated for individual patients, regardless of dose level. Descriptive statistics will be used to summarize PSA, and changes in it. Serial PSA levels will be displayed using spaghetti plots, and changes in PSA using waterfall plots.
Change TAM levels as measured by immunohistochemistry | Baseline to month 2
  Frequency distributions will be generated for patients treated at the MTD. Descriptive statistics will be used to summarize all markers, and changes in them.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth I. Heath, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (3):
- United States (3):
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute at McLaren Northern Michigan - Petoskey Radiation Oncology, Petoskey, Michigan
  - Karmanos Cancer Institute at McLaren Northern Michigan- Petoskey Medical Oncology, Petoskey, Michigan